CLINICAL TRIAL: NCT00768170
Title: A Open-Label, Single Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of MK0633 in Japanese Asthmatic Children Aged 12 to Less Than 16 Years
Brief Title: MK0633 Single Dose Study in Japanese Asthmatic Children Aged 12 to Less Than 16 Years (0633-028)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0633-028; MK0633-028; 2008_552
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — MK-0633 p-toluenesulfonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MK0633
  Interventions: Drug: MK0633

INTERVENTIONS:
Drug: MK0633 — MK0633 (50 mg) Oral, single dose

SUMMARY:
This study evaluates the safety, tolerability and pharmacokinetics (PK) of MK0633 in adolescent mild-to-moderate Japanese asthma patients to permit further clinical investigation

ELIGIBILITY:
Inclusion Criteria:

* Patient Is Judged To Be In Good Health, Other Than Having Mild To Moderate Asthma, Based On Medical History, Physical Examination, Vital Signs, And Laboratory Safety Tests
* Patient Has No Clinically Significant Abnormality On Electrocardiogram (Ecg) Performed At The Prestudy (Screening) Visit And/Or Prior To Administration Of The Initial Dose Of Study Drug
* Patient Has At Least 1 Year Of Mild-To-Moderate Asthma
* Patient Has Been A Nonsmoker For At Least 6 Months
* Patients Of Childbearing Potential Must Agree To Use A Medically Acceptable Method Of Contraception During The Study
* Patients Must Be Able To Swallow Tablets

Exclusion Criteria:

* Patient Has A History Of Clinically Significant Endocrine, Gastrointestinal, Cardiovascular, Hematological, Hepatic, Immunological, Renal, Respiratory, Other Than Asthma, Or Genitourinary Abnormalities Or Diseases
* Patient Has Required A Visit To A Hospital Or Emergency Room Due To An Asthma Exacerbation Within 3 Months Of The Prestudy Visit
* Patient Has Unresolved Signs And Symptoms Of An Upper Respiratory Tract Infection (Uri) Or Has Had Had An Upper Respiratory Tract Infection Within 3 Weeks Prior To The Prestudy Visit
* Patient Has A History Of Stroke, Chronic Seizures, Or Major Neurological Disorder
* Patient Has A History Of Neoplastic Disease
* Use Of Theophylline, Anti-Allergic Compounds (Except For Nasal Drop And Eye-Drop Omalizumab, Zileuton, Oral Corticosteroid, And Oral Beta Agonists (Including Patch) Are Excluded ~ 2 Weeks Prior To Administration Of Study Drug And Throughout The Study 7)Patient Consumes Alcoholic Beverages

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of MK0633 in adolescent asthma patients based on any clinical or laboratory adverse experiences | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC